CLINICAL TRIAL: NCT03781206
Title: Efficacy of Negative Pressure Wound Therapy (NPWT) for Prevention of Wound Infection and Improvement of Wound Healing After Stoma Reversal
Brief Title: Negative Pressure Wound Therapy for Wound Healing After Stoma Reversal
Acronym: NESTOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 824
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Stoma Site Infection
Keywords: Stoma; Surgical Site Infection; Negative Pressure Wound Therapy
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): After stoma reversal, patients of SOC group will be treated as for normal clinical practice, using a simple adhesive wound dressing.
- Negative Pressure Wound Therapy (NPWT) (Experimental): PICO™ 7 will be applied after stoma reversal
  Interventions: Device: PICO™ 7

INTERVENTIONS:
Device: PICO™ 7 — PICO™ system (Smith&Nephew Healthcare, Hull, UK) is a Single-Use Negative Pressure Wound Therapy (NPWT) System consisting of a small portable pump, 2 lithium batteries, 2 dressings and fixation strips.
  Arms: Negative Pressure Wound Therapy (NPWT)

SUMMARY:
Stoma reversal is associated with high incidence of post-surgical complications, including Surgical Site Infections (SSI). Negative Pressure Wound Therapy (NPWT) has been successfully applied to surgical wound management, reducing the SSIs incidence. This is a randomized open-label trial to assess the efficacy of NPWT in decreasing the rate of SSI after stoma reversal.

DETAILED DESCRIPTION:
Stoma reversal after abdominal resection is associated with several complications, of which the most common is wound infection. Surgical Site Infections (SSI) usually result in increased long-term complications, such as incisional hernia, prolonged hospital stay, increased outpatients visits and medical costs. Negative-Pressure-Wound-Therapy (NPWT) is a technique using vacuum dressing, commonly used to promote surgical wound healing, but there is a significant lack of knowledge about its safety and efficacy in promoting wound healing after stoma closure. This is an interventional, randomized, open label trial to evaluate the safety and efficacy of the NPWT (PICO™ system, Smith&Nephew Healthcare, Hull, UK) on stoma wound compared to Standard of Care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, any sex;
* Patients who underwent elective open or laparoscopic rectal resection ostomy construction (loop/end ileostomy; loop/end colostomy) for either oncological and Inflammatory Bowel Disease (IBD) indications;
* Normal water contrast enema prior to surgery;
* Both neo-adjuvant and adjuvant treatment are allowed for cancer patients;
* Both immunosuppressant and biological medications are allowed for IBD patients.

Exclusion Criteria:

* Patients age at screening < 18 years;
* Pregnant or breastfeeding women;
* Neurodegenerative disorders or psychiatric diseases;
* Contraindications or hypersensitivity to the use of the investigational product or its components;
* Patients with skin features (e.g., tattoos, pre-existing scarring) which could interfere with the study assessments;
* Patients with post-operative bleeding (to be assessed 24 hours after surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) rate comparison | Post-operative day 7
  The rate of superficial (infections involving only the skin and subcutaneous tissue) or deep (infections involving the muscle and the fascia but not organ space) SSI will be assessed by medical examination
Surgical Site Infection (SSI) rate comparison | Post-operative day 30
  The rate of superficial (infections involving only the skin and subcutaneous tissue) or deep (infections involving the muscle and the fascia but not organ space) SSI will be assessed by medical examination

SECONDARY OUTCOMES:
Wound healing timing comparison | Post-operative day 30
  Wound healing is defined as complete tissue restoration, scar formation and absence of resected tissues and will be assessed by medical examination
Quality of life assessment | Post-operative day 7
  Quality of life will be assessed using the EuroQol-5 Dimension-5 Levels (EQ5D5L) questionnaire. The EQ5D5L questionnaire comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The questionnaire also includes a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Quality of life assessment | Post-operative day 30
  Quality of life will be assessed using the EuroQol-5 Dimension-5 Levels (EQ5D5L) questionnaire. The EQ5D5L questionnaire comprises 5 dimensions (mobility, self) care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The questionnaire also includes a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Quality of life assessment | Post-operative day 90
  Quality of life will be assessed using the EuroQol-5 Dimension-5 Levels (EQ5D5L) questionnaire. The EQ5D5L questionnaire comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The questionnaire also includes a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Quality of life assessment | Post-operative day 180
  Quality of life will be assessed using the EuroQol-5 Dimension-5 Levels (EQ5D5L) questionnaire. The EQ5D5L questionnaire comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The questionnaire also includes a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Pain assessment | Post-operative day 7
  Pain will be measured using the McGill Pain questionnaire. The questionnaire presents a list of 78 words in 20 sections that are related to pain. The users mark the words that best describe their pain (multiple markings are allowed). Among the words, sections of these words signify different components of pain: Sensory (sections 1-10), Affective (sections 11-15), Evaluative (section 16), and Miscellaneous (sections 17-20).
Pain assessment | Post-operative day 30
  Pain will be measured using the McGill Pain questionnaire. The questionnaire presents a list of 78 words in 20 sections that are related to pain. The users mark the words that best describe their pain (multiple markings are allowed). Among the words, sections of these words signify different components of pain: Sensory (sections 1-10), Affective (sections 11-15), Evaluative (section 16), and Miscellaneous (sections 17-20).
Pain assessment | Post-operative day 90
  Pain will be measured using the McGill Pain questionnaire. The questionnaire presents a list of 78 words in 20 sections that are related to pain. The users mark the words that best describe their pain (multiple markings are allowed). Among the words, sections of these words signify different components of pain: Sensory (sections 1-10), Affective (sections 11-15), Evaluative (section 16), and Miscellaneous (sections 17-20).
Pain assessment | Post-operative day 180
  Pain will be measured using the McGill Pain questionnaire. The questionnaire presents a list of 78 words in 20 sections that are related to pain. The users mark the words that best describe their pain (multiple markings are allowed). Among the words, sections of these words signify different components of pain: Sensory (sections 1-10), Affective (sections 11-15), Evaluative (section 16), and Miscellaneous (sections 17-20).

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No